CLINICAL TRIAL: NCT01202162
Title: A Comparison of Desflurane vs. Sevoflurane on Time to Awakening and the Incidence and Severity of Cough After Ambulatory Surgery Using Laryngeal Mask Airway
Brief Title: A Comparison of Desflurane vs. Sevoflurane and the Time to Awakening and the Incidence and Severity of Cough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Gildasio De Oliveira, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: STU00036200
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Results first posted 2013-07-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-10

CONDITIONS: Surgery; Anesthesia
Keywords: Induction; Coughing; Anesthesia
MeSH Terms: conditions — Cough | interventions — Desflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desflurane (Active Comparator): Administration of Desflurane
  Interventions: Drug: Desflurane
- Sevoflurane (Active Comparator): Administration of Sevoflurane
  Interventions: Drug: Administration of Sevoflurane

INTERVENTIONS:
Drug: Desflurane — Administratino of Desflurane
  Arms: Desflurane
Drug: Administration of Sevoflurane — Administration of Sevoflurane
  Arms: Sevoflurane

SUMMARY:
Goals for ambulatory surgery include providing optimal surgical conditions while ensuring a rapid early recovery without side effect. Dexter et al1 concluded in a meta-analysis that Desflurane can reduce the extubation time when compared to Sevoflurane. This potential benefit of Desflurane can be especially attractive in short ambulatory cases performed with general anesthesia with a laryngeal mask airway.

Although some studies have not shown a difference on perioperative cough and laryngospasm between Desflurane and Sevoflurane at clinically relevant doses.It has been reported in the literature that Desflurane causes cough4 and many providers avoid using Desflurane with a LMA (laryngeal mask airway) in the ambulatory setting. In this study we will also evaluate, as a secondary outcome, the presence and severity of perioperative cough and laryngospasm.

Previous investigators have demonstrated a more rapid resumption of normal daily activities after ambulatory surgery in patients anesthetized with Desflurane when compared with Sevoflurane.these investigators suggested a better quality of recovery when Desflurane is used probably due to a lower lipid solubility of Desflurane. We will also evaluate quality of recovery as a secondary outcome using a validated instrument.

Significance:

1. A more rapid awakening, especially, in a fast and high turnover cases that are performed with LMA can lead to a more cost effective utilization of operating room time
2. It has been reported that Desflurane causes more cough than Sevoflurane and Anesthesiologists avoid using Desflurane with LMA cases, this study will reinforce that there is no difference.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Female patients undergoing outpatient gynecologic and breast surgery
* Under general anesthesia using an LMA
* ASA I,II,

Exclusion Criteria:

* Patients on CNS depressants
* Chronic opioid use
* Corticosteroid
* Pregnant patients
* Full stomach
* Morbidly obese (BMI >35kg/m2)
* Hepatitis B
* Hepatitis C
* Coronary artery disease
* Liver disease
* Renal disease
* Seizure disorder

Dropout criteria:

* Need for endotracheal tube
* Surgeon or patient request
* Hospital admission

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2010-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gildasio De Oliveira, M.D, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Dexter F, Bayman EO, Epstein RH. Statistical modeling of average and variability of time to extubation for meta-analysis comparing desflurane to sevoflurane. Anesth Analg. 2010 Feb 1;110(2):570-80. doi: 10.1213/ANE.0b013e3181b5dcb7. Epub 2009 Oct 9. PMID 19820242
- [Background] McKay RE, Bostrom A, Balea MC, McKay WR. Airway responses during desflurane versus sevoflurane administration via a laryngeal mask airway in smokers. Anesth Analg. 2006 Nov;103(5):1147-54. doi: 10.1213/01.ane.0000237293.39466.65. PMID 17056947
- [Background] White PF, Eshima RW, Maurer A, King T, Lin BK, Heavner JE, Bogetz MS, Kaye AD. A comparison of airway responses during desflurane and sevoflurane administration via a laryngeal mask airway for maintenance of anesthesia. Anesth Analg. 2003 Mar;96(3):701-705. doi: 10.1213/01.ANE.0000048978.40522.AB. PMID 12598249
- [Background] Arain SR, Shankar H, Ebert TJ. Desflurane enhances reactivity during the use of the laryngeal mask airway. Anesthesiology. 2005 Sep;103(3):495-9. doi: 10.1097/00000542-200509000-00011. PMID 16129973
- [Background] Mahmoud NA, Rose DJ, Laurence AS. Desflurane or sevoflurane for gynaecological day-case anaesthesia with spontaneous respiration? Anaesthesia. 2001 Feb;56(2):171-4. doi: 10.1046/j.1365-2044.2001.01528.x. PMID 11167479

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 85 Subjects were recruited and randomized and 80 completed the study. Subjects were consecutively enrolled from December 2010 through February 2012.
Period: Overall Study
Arm/Group | Desflurane | Sevoflurane
Started | 43 | 42
Completed | 40 (40 completed the intraoperative through discharge phase of the study.) | 40 (40 completed the intraoperative through discharge phase of the study.)
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desflurane | Sevoflurane | Total
Number analyzed (Participants) | 43 | 42 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 42 | 85
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.2 (8.3) | 39.9 (7.7) | 40.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 42 | 85
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 43 | 42 | 85

OUTCOME MEASURES:

1. Primary Outcome: Time to Awakening
Time Frame: Time inhalational agent is turned off to time of patient awakening
Measure: Median (Inter-Quartile Range); unit: Elapsed time in minutes
Arm/Group | Desflurane | Sevoflurane
Number analyzed (Participants) | 40 | 40
Elapsed time in minutes | 6.8 [5.0 to 9.6] | 11.8 [8.8 to 14.6]

2. Secondary Outcome: Number of Participants Who Coughed
Time Frame: Perioperative
Measure: Number; unit: participants
Arm/Group | Desflurane | Sevoflurane
Number analyzed (Participants) | 40 | 40
participants | 4 | 7

3. Secondary Outcome: Quality of Recovery 40
Description: Survey completion at 24 hours post surgery of the Quality of Recovery 40 questionnaire.This questionnaire asks 40 questions in 5 categories of recovery. The scores are combined from each group and are used as a composite score. The scores range from a low of 40 to a high of 200. A score of 40 would indicate a poor quality of recovery where as a score of 200 would be a good quality of recovery at 24 hours postoperative.
Time Frame: 1 day
Population: In the Desflurane group 35 completed the survey 24 hours postoperative where as 33 in the Sevoflurane completed the survey during the postoperative period.
Measure: Median (Inter-Quartile Range); unit: score (between 40 low-200 high)
Arm/Group | Desflurane | Sevoflurane
Number analyzed (Participants) | 35 | 33
score (between 40 low-200 high) | 188 [185 to 191] | 182 [176 to 190]

ADVERSE EVENTS:
Time Frame: Intraoperative period from induction of anesthesia until time of discharge from the operating room.
Description: Laryngospasm occuring from the introduction of inhalation agent to time of discharge from the operating room
Arm/Group | Desflurane | Sevoflurane
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 2/40 | 1/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Desflurane (N=40) | Sevoflurane (N=40)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 2/38 (2) | 1/39 (1)

LIMITATIONS AND CAVEATS:
Our study is only valid if interpreted within the context of its limitations. We have only evaluated female subjects undergoing ambulatory hysteroscopic surgery which limits the generalizability of our results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No